CLINICAL TRIAL: NCT07274137
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of MDR-001 Administered Orally Over 52 Weeks in Participants With Overweight or Obesity (MOBILE)
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of MDR-001 in Adult Participants With Overweight or Obesity (MOBILE）
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MindRank AI Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDR-001-CN-05
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MDR-001 Dose 1 (Experimental)
  Interventions: Drug: MDR-001
- MDR-001 Dose 2 (Experimental)
  Interventions: Drug: MDR-001
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDR-001 — Participants will Receive Small Molecule MDR-001 Tablets Administered Orally
  Arms: MDR-001 Dose 1; MDR-001 Dose 2
Drug: Placebo — Participants will Receive Placebo
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, phase III clinical study to evaluate the efficacy and safety of the oral small molecule MDR-001 Tablets over 52 weeks as an adjunct to a lifestyle intervention in participants with overweight or obesity.The goal of this clinical trial is to determine whether the oral drug MDR-001 can improve weight management in adult participants with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate in this study
* Chinese male or female participants who are aged 18-65 (inclusive) years at the time of signing the ICF
* Participants who are obesity (BMI ≥ 28.0 kg/m2), or overweight (24.0 kg/m2 ≤ BMI < 28.0 kg/m2) with at least one of the the following weight-related comorbidities at screening:1) Pre-diabetes. 2) Hypertension.3) Dyslipidemia.4) Fatty liver.5) Obstructive sleep apnea syndrome.6) Complaint of weight-bearing joint pain.
* Participants had a stable weight maintenance during the 3 months of dietary and physical activity prior to screening (participant-reported data acceptable) and no more than 5% weight fluctuation

Exclusion Criteria:

* Obesity induced by secondary diseases or drug
* Have diabetes mellitus
* Have any lifetime history of a suicidal attempt or suicidal behavior
* Have a history of depressive disorder
* History of gout within 6 months prior to screening
* History of major cardiovascular or cerebrovascular disease within 6 months prior to screening, defined as:1)Acute myocardial infarction (MI), percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), heart valve repair/replacement, unstable angina, hemorrhagic stroke (stroke), ischemic stroke (including transient ischemic attack [TIA]).2)Congestive heart failure of New York Heart Association (NYHA) class III or IV.3)Severe arrhythmias
* History of malignancy within 5 years prior to screening or newly diagnosed malignancy at screening
* Have a family or personal history (parents, children, and siblings of medullary thyroid cancer or Multiple Endocrine Neoplasia Syndrome Type 2 .
* Abnormal thyroid function tests at screening not adequately controlled by stable medication doses , or thyroid ultrasound at screening showing thyroid nodules classified as Chinese-thyroid imaging-reporting and data system category 4 or higher.
* History of significant gastrointestinal disease or gastrointestinal surgery or clinically significant gastric emptying abnormality within 6 months prior to screening.
* History of intestinal disorders deemed clinically significant by the investigator, or acute hemorrhoidal episode within 3 months prior to screening.
* History of acute or chronic pancreatitis, or abnormally elevated serum amylase or lipase levels at screening.
* revious acute or chronic hepatitis, or symptoms and signs of any other liver disease other than non-alcoholic fatty liver disease, or abnormalities in related laboratory tests at screening
* Presence of acute or chronic cholecystitis at screening, or symptomatic or treatment-requiring cholelithiasis/gallbladder polyps at screening, or newly diagnosed cholelithiasis within 6 months before screening
* Hypersensitivity or suspected hypersensitivity to glucagon-like peptide 1 receptor agonist (GLP-1RA) drugs or excipients.
* History of drug abuse or dependence prior to screening.
* Have current or history of treatment with medications that may cause significant weight gain within 3 months prior to screening, including but not limited to:

  1. Approved/unapproved marketed weight-loss drugs: orlistat, sibutramine hydrochloride, phentermine, phentermine-topiramate, naltrexone-amfebutamone, tirzepatide, semaglutide, liraglutide, beinaglutide, phendimetrazine, methylamphetamine, etc.
  2. Investigational products of weight-loss: Glucagon-like peptide 1 receptor (GLP-1R) agonists, GLP-1R/glucagon receptor (GCGR) agonists, glucose-dependent insulinotropic polypeptide receptor (GIPR)/GLP-1R agonists, GIPR/GLP-1R/GCGR agonists,GLP-1R agonists/activin type II receptor (ActRII) inhibitors, GLP-1R/GIPR/fibroblast growth factor 21 receptor (FGF21R) agonists or FGF21R/GCGR/GLP-1R agonists.
  3. Hypoglycemic drugs, such as metformin, sodium-glucose cotransporter 2 (SGLT2) inhibitors, thiazolidinediones (TZDs) or dipeptidyl peptidase 4 (DPP-4) inhibitors.
  4. Systemic steroid therapy (including intravenous, oral, intra-articular).
  5. Tricyclic antidepressants or other antipsychotic or antiepileptic drugs affecting body weight (e.g., mirtazapine, paroxetine, clozapine, olanzapine, risperidone, quetiapine, paliperidone, valproic acid, valproic acid derivatives, lithium).
* History of bariatric surgery (excluding acupuncture/cupping/catgut embedding for bariatric surgery, liposuction, and abdominoplasty performed >1 year prior to screening) or plans to undergo bariatric surgery or acupuncture/cupping/catgut embedding, liposuction, abdominoplasty during the study period.
* Planned chronic use of medications affecting gastrointestinal motility or scheduled gastric emptying-impairing surgery during the study period.
* Major or medium-sized surgery, or severe trauma or serious infection within 3 months prior to screening, which, as assessed by the investigator, would preclude trial participation, or planned surgery during the study period (excluding outpatient procedures deemed by the investigator to have no impact on subject safety or trial outcomes).
* History of organ transplant.
* Use of any drug or food known to potently or moderately inhibit or induce cytochrome P450 3A4 enzyme (CYP3A4) and/or inhibit P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study.
* Currently participating in any other clinical study, or if received any investigational product or medical devices within ≤ 3 months or 5 half-lives (t1/2) prior to screening, whichever is longer.
* Donation or loss of ≥ 400 mL of blood or transfusion/blood products during this period within 3 months prior to screening, or intention to donate blood during the study.
* emale participants during pregnancy or lactation.
* The investigator, site personnel, and/or their immediate family members directly related to the study. An immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Participants who may be unable to complete this study for other reasons, or have other conditions that, as assessed by the investigator, will make the participant unsuitable for participation in this study, for example, the participant refuses to use only the weight-loss drugs specified in the protocol during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in body weight (%) at Week 52 | baseline,Week 52
  (Week 52 body weight-baseline body weight)/baseline weight
Percentage (%) of participants who achieve≥5% body weight reduction from baseline at Week 52 | baseline,Week 52
  (Week 52 body weight-baseline body weight)/baseline body weight, who achieve≥5%

SECONDARY OUTCOMES:
Change from baseline in body weight (kg) at Week 52 | baseline,Week 52
  Week 52 body weight-baseline body weight
Percentage (%) of participants who achieve ≥ 10% or ≥ 15% body weight reduction from baseline at Week 52 | Baseline,Week52
  (Week 52 body weight-baseline body weight)/baseline body weight, who achieve≥ 10% or ≥ 15%
Change from baseline in BMI (kg/m2) at Week 52 | Baseline,Week52
  BMI (kg/m2) = weight (kg)/height (m)2
Change from baseline in waist circumference (cm) at Week 52 | Baseline, Week52
  Week 52 waist circumference-baseline waist circumference
Change from baseline in hip circumference (cm) at Week 52 | Baseline,Week 52
  Week 52 hip circumference-baseline hip circumference
Change from baseline in waist-hip ratio (%) at Week 52 | Baseline,Week52
  Waist-to-hip ratio = waist circumference (cm) / hip circumference (cm)
Change from baseline in Total cholesterol (TC, mmol/L) at Week 52 | Baseline, Week 52
  Week 52 Total cholesterol-baseline Total cholesterol
Change from baseline in Triglycerides (TG, mmol/L) at Week 52 | baseline,Week 52
  Week 52 Triglycerides-baseline Triglycerides
Change from baseline in Low-density lipoprotein cholesterol (LDL-C, mmol/L) at Week 52 | baseline,Week 52
  Week 52 Low-density lipoprotein cholesterol-baseline Low-density lipoprotein cholesterol
Change from baseline in High-density lipoprotein cholesterol (HDL-C，mmol/L) at Week 52 | baseline,Week 52
  Week 52 High-density lipoprotein cholesterol-baseline High-density lipoprotein cholesterol
Change from baseline in Non-high-density lipoprotein cholesterol (nHDL-C, mmol/L) at Week 52 | baseline,Week 52
  Week 52 Non-high-density lipoprotein cholesterol-baseline Non-high-density lipoprotein cholesterol
Change from baseline in Lipoprotein (a) (Lp[a], mg/dL) at Week 52 | baseline，Week 52
  Week 52 Lipoprotein -baseline Lipoprotein
Change from baseline in Systolic blood pressure (SBP, mmHg) at Week 52 | baseline，Week 52
  Week 52 Systolic blood pressure-baseline Systolic blood pressure
Change from baseline in Diastolic blood pressure (DBP, mmHg) at Week 52 | baseline，Week 52
  Week 52 Diastolic blood pressure-baseline Diastolic blood pressure
Change from baseline in Glycosylated hemoglobin (HbA1c, %) at Week 52 | baseline，Week 52
  Week 52 Glycosylated hemoglobin-baseline Glycosylated hemoglobin
Change from baseline in Fasting plasma glucose (FPG, mmol/L) at Week 52 | baseline，Week 52
  Week 52 Fasting plasma glucose-baseline Fasting plasma glucose
Adverse events | baseline，Week 52
  Number of participants with treatment-related adverse events as assessed by mild, moderate and severe

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - Peking University People's Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - People's Hospital of Hunan Province, Changsha
  - The Fourth Hospital of Changsha, Changsha
  - The Third People's Hospital of Datong, Datong
  - Dongyang People's Hospital, Dongyang
  - Ganzhou People's Hospital, Ganzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - The SecondPeople's Hospital of Hefei, Hefei
  - Huizhou Central People's Hospital, Huizhou
  - Huizhou Third People's Hospital, Huizhou
  - Huzhou Central Hospital, Huzhou
  - Central Hospital Affiliated To Shangdong First Medical University, Jinan
  - Central Hospital of Jin zhou, Jinzhou
  - Jingzhou Hospital Affiliated to Yangtze University, Jinzhou
  - The Third Affiliated Hospital of Jinzhou Medical University, Jinzhou
  - JiuJiang No.1 people's Hospital, Jiujiang
  - Lianyungang Hospital of TCM, Lianyungang
  - Liaocheng People's Hospital, Liaocheng
  - Loudi Central Hospital, Loudi
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - Sanya Central Hospital (Hainan Third People's Hospital), Sanya
  - Shenyang Fifth People Hospital, Shenyang
  - Shenyang Sixth People's Hospital, Shenyang
  - The People's Hospital of liaoning Province, Shenyang
  - The Second Hospital of Hebei Medical University, Shijia Zhuang
  - Siping Central People's Hospital, Siping
  - The First Affiliated Hospital of Soochow University, Suzhou
  - First Hospital of Shanxi Medical University, Taiyuan
  - Shanxi Bethune Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang province, Taizhou
  - Wuhan Third Hospital•Tongren Hospital of Wuhan University, Wuhan
  - Xuancheng People's Hospital, Xuancheng
  - Yichang Central People's Hospital, Yibin
  - Yichang Central People's Hospital, Yichang
  - Yueyang Central Hospital, Yueyang
  - Yueyang People's Hospital, Yueyang
  - The Second Affiliated Hospital of ZhengzhouUniversity, Zhengzhou
  - The Third People's Hospital of Zhengzhou, Zhengzhou
  - Xiangya Hospital Zhuzhou Central South University, Zhuzhou
  - PKUCare Luzhong Hospital, Zibo
  - Zibo Central Hospital, Zibo
  - Zibo Municipal Hospital, Zibo